CLINICAL TRIAL: NCT02071043
Title: Trial of Xeloda and Oxaliplatin (XELOX) as Neo-adjuvant Chemotherapy Followed by Surgery in Advanced Gastric Cancer Patients With Para-aortic Lymph Node Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-ON-03
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Gastric Cancer
Keywords: neo-adjuvant chemotherapy; advanced gastric cancer patients; para-aortic lymph node metastasis
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XELOX (Experimental): XELOX: Schedule of Oxaliplatin plus capecitabine (XELOX) will be as follow:
  Capecitabine 1000 mg/m2 ，orally taken 30 minutes after meal, bid ， d 1~14 every 3 weeks(treatment for 2 weeks and rest 1 week) Oxaliplatin：130mg/m2， iv infusion over 2h，d1,every 3 weeks
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000 mg/m2 ，orally taken 30 minutes after meal, bid ， d 1~14 every 3
Drug: Oxaliplatin — Oxaliplatin：130mg/m2， iv infusion over 2h，d1,every 3 weeks

SUMMARY:
Gastric cancer with para-aortic lymph node (PAN) involvement is regarded as advanced disease, and only chemotherapy is recommended from the guidelines. In unresectable cases, neoadjuvant chemotherapy could prolong survival if conversion to resectability could be achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric or gastroesophageal adenocarcinoma proven histologically .
2. Has para-aortic lymph node metastasis(PAN was defined as nodes in the region between the upper margin of the celiac artery and the upper border of the inferior mesenteric artery (stations no. 16a2/16b1))
3. Eastern Cooperative Oncology Group performance status of 0 to 1.
4. Life expectancy ≥12 weeks.
5. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).

   Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN , ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L。 Adequate renal function: Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
6. Female subjects should not be pregnant or breast-feeding.
7. No serious concomitant disease that will threaten the survival of patients to less than 5 years.

Exclusion Criteria:

1. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
2. History of another malignancy in the last 5 years with the exception of the following:

   Any previous palliative, adjuvant or neoadjuvant chemotherapy and/or radiotherapy. Prior treatment for locally advanced or metastatic gastric cancer.
3. Any other metastatic disease will render patient ineligible according to AJCC staging manual(such as liver，lung，etc）.
4. Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
5. Poorly controlled diabetes mellitus with fasting blood sugar > 18 mm. Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
6. Unstable, persistent cardiac disease despite medicinal treatment, myocardial infarction within 6 months before the start of the trial
7. Previous surgery on primary tumour; Prior palliative surgery (open and closure, passage operation)
8. Any other type of tumour (e.g. leiomyosarcoma, lymphoma) or a secondary malignancy, excepting basal cell skin carcinoma or basal cell carcinoma in situ of the cervix which have already been successfully treated -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The primary study end point was the response rate of preoperative XELOX followed by surgery in gastric cancer patients with PAN involvement | 8 Months after the last subject participate in
  evaluation will be based on tumor assessment with follow-up, including chest and upper-abdominal During preoperative treatment period, CT scan will be performed every 6 -8 weeks (2 cycles after).After surgery, CT scan will be planned every 3 months, brain MRI and bone scan (ECT) will be performed if any suspected symptoms occur.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 40 Months after the last subject participate in
  be based on tumor assessment with follow-up, including chest and upper-abdominal During preoperative treatment period, CT scan will be performed every 6 -8 weeks (2 cycles after).After surgery, CT scan will be planned every 3 months, brain MRI and bone scan (ECT) will be performed if any suspected symptoms occur.
overall survival | 3 years after the last subject participate in
  out-patient clinic and telephone visit will be done every 3 months for the first two years, and every 6 months after two years
Grade 3 or 4 Adverse Events as a Measure of Safety | 1 year after the last subject finish the treatment
  Adverse Events will measure in the whole study according to CTC-AE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, Doctor, Principal Investigator — Medicine-Oncology Derpartment of Zhongshan hospital
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China